CLINICAL TRIAL: NCT00851656
Title: MilkScreen Home Test for Alcohol in Breast Milk Clinical Study
Brief Title: MilkScreen Home Test for Alcohol in Breast Milk
Status: Completed | Type: Observational
Sponsor: UpSpring Baby, Ltd. (Industry)
Responsible Party: Julie Jumonville, Chief Product Officer, UpSpring, Ltd.
Other Study IDs: 4001-001
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Alcohol Concentrations in Body Fluids

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the performance of the UpSpring Milkscreen Test for Alcohol in Breast Milk to detect alcohol in breast milk from lactating women.

DETAILED DESCRIPTION:
The Milkscreen Test for alcohol in Breast Milk is intended for use by lactating mothers as a rapid qualitative detection for the presence of alcohol in their breast milk prior to offering the breast milk to their nursing infant. This study will obtain data to demonstrate the sensitivity and specificity of MilkScreen™ compared to the reference method, Gas Chromatography (GC) for alcohol content and will additionally provide validation of the usability of the device by for over-the-counter use.

The study will enroll approximately 50 lactating mothers who will come into a center in small groups in a contrived social setting like a wine tasting. Upon completion of informed consent and demonstration of meeting inclusion/exclusion criteria, subjects will be tested with disposable breathalyzer test and baseline breast milk samples provided. The baseline breast milk samples will be tested with the test article by the subject. Aliquots from the same samples will be prepared for testing by an outside lab with GC and with the test article.

Subjects will be asked to provide baseline demographics such as height and weight, days since birth of child, race/ethnicity, and information about any prescription or OTC drugs, herbal compounds or vitamins they have taken in the previous 72 hours.

Subjects will be provided with up to 3 standard alcohol drinks over the course of a two hour period. At prescribed time intervals following consumption, subjects will be asked to provide a breast milk sample and to submit to a breathalyzer test. Each breast milk sample will be tested by the subject with the test article following the labeling instructions only and the sample will also be aliquoted into tightly sealing, low head space samples containers for method comparison testing by an outside lab on GC and again with MilkScreen™.

Subjects will be asked to drink at least one drink, but may ingest up to two additional alcoholic beverages. Each subject's intoxication state will be monitored before each additional drink is provided and will not be allowed to consume additional drinks if their BAC as measured by the disposable breathalyzer device exceeds 0.10% (100 mg/dL). All drinks will be measured for consistency and subjects will be asked to self report whether they finished their drink at the point when samples are taken. Subjects will be provided with transportation using designated non-drinking drivers.

Samples of breast milk taken both prior to and following the ingestion of alcohol will be coded and thereby blinded to the lab. The lab will run both GC and MilkScreen™ testing on each sample and report the results as paired. This data will be analyzed to demonstrate that the MilkScreen™ Home Test for Alcohol in Breast Milk has sufficient sensitivity and specificity as compared to the reference method, GC, to support the test article's intended use.

Subjects will be asked to complete a questionnaire on the usability of the labeling instructions on MilkScreen™ Home Test for Alcohol in Breast Milk to demonstrate that consumers can use the directions properly to test their breast milk for the presence of alcohol and properly interpret the results.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age equal to or greater than 21 years
* Actively breast-feeding
* Willing to drink at least one alcoholic beverage (wine or beer) during study in a controlled setting
* Willing to arrive to the study session prior to consuming any alcoholic beverages within the last 6 hours.
* Willing to attend single session study for 3-4 hours duration until their BAC drops below 0.06%
* Willing to accept designated driver or study-supplied transportation
* Willing to agree to not breast feed their infant for 2 hour following leaving the study session
* English language fluency

Exclusion Criteria:

* Distance of more than 25 miles from study site
* Pregnant (hCG test will be administered prior to alcohol consumption)
* Communicable diseases (e.g., Flu)
* HIV Positive
* History of Alcoholism (Recorded on the CRF)
* Arriving to the study session with a BAC at or below 0.01%
* Any medical condition which precludes the subject from drinking alcohol

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lactating women, 21 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zeis Consulting Group, San Marcos, California, United States